CLINICAL TRIAL: NCT05577689
Title: Combining Multi-omics Analysis and Organoid Models to Search for Novel Therapy Target in Metastatic Prostate Cancer
Brief Title: Novel Therapy Target in Metastatic Prostate Cancer
Acronym: NTTPro
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ding-Wei Ye, Fudan University Shanghai Cancer Center, Fudan University
Other Study IDs: PCa-Organoid
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Prostate Neoplasms
Keywords: prostate cancer; multi-omics; organoid
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Histocompatibility Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients: There is only one arm in the trial
  Interventions: Other: Tissue

INTERVENTIONS:
Other: Tissue — Tissue will be derived from patients during a standard of care procedure

SUMMARY:
The aim of this study is to use multiomics sequencing to explore the molecular characteristics of metastatic prostate cancer (mPCa), especially metastatic castration-resistant prostate cancer (mCRPC). At the same time, mCRPC models will be constructed, including organoids and animal models, serving as a basic and translational research platform to help identify novel drug targets for mPCa.

DETAILED DESCRIPTION:
Although substantial progress in treatments for prostate cancer have been made in the past decades, distant metastasis and drug resistance remained a major cause of prostate cancer-related deaths. The five-year survival rate for men with mPCa was only 30% and all patients with mPCa would inevitably progress to the castration-resistant stage with limited therapeutic chance. In China, the current situation is more worrying, with rapidly increasing PCa incidence and higher proportion of mPCa diagnosed compared with the Western nations (~30% vs ~5%).

Multiomics sequencing provides a promising strategy to discover the underlying molecular basis driving metastasis and resistance and identify the new treatment strategies for patients with mCRPC. The candidate drug target revealed by the multiomics sequencing could be further examined in the organoid and animal models, facilitating the clinical application from basic discovery.

This study can establish a mCRPC research system to find the molecular mechanism and potential intervention targets of mCRPC, thereby paving the way for the discovery of new treatments for mCRPC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed prostate cancer
2. metastatic disease confirmed by image examination
3. Patients who can undergo surgery or biopsy for prostate cancer
4. Able to provide informed consent

Exclusion Criteria:

1. Patients diagnosed with other types of cancer besides prostate cancer
2. Not accessible to surgery sample
3. Patients fail to provide informed consent
4. Other situation that researchers think are unsuitable for this study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic prostate cancer especially metastatic castration resistant prostate cancer will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Multiple omics features | 3 years
  Multi-omics information including genetic profiling results, transcriptional profiling results and epigenomic profiling results will be collected and analyzed.
Organoids successfully generated from metastatic prostate cancer | 3 years
  Successful isolation of prostate cancer organoids from surgical specimens of patients diagnosed with metastatic prostate cancer. We will calculate the culture efficiency and total number of organoids generated in our center.
Developing of biomarkers related to cancer metastasis and drug resistant | 3 years
  To search for biomarkers related to tumor metastasis and resistance by performing multi-omics analysis to surgery specimens derived from patients with metastatic prostate cancer.

SECONDARY OUTCOMES:
Animal models successfully generated from patient derived prostate cancer organoids | 3 years
  Prostate cancer organoids with clarified characteristics will be transplanted into mice to establish PDOX models.
Response of the prostate cancer organoids to the selected anti-cancer compounds | 3 years
  Organoid that are successfully cultured and characteristic clarified will be treated with the selected compounds to test their anti-cancer activity.
Response of the PDOX models to the selected anti-cancer compounds | 3 years
  PDOX models that successfully established will be treated with the selected compounds to test their anti-cancer activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akhoundova D, Rubin MA. Clinical application of advanced multi-omics tumor profiling: Shaping precision oncology of the future. Cancer Cell. 2022 Sep 12;40(9):920-938. doi: 10.1016/j.ccell.2022.08.011. Epub 2022 Sep 1. PMID 36055231
- [Background] Yerly L, Pich-Bavastro C, Di Domizio J, Wyss T, Tissot-Renaud S, Cangkrama M, Gilliet M, Werner S, Kuonen F. Integrated multi-omics reveals cellular and molecular interactions governing the invasive niche of basal cell carcinoma. Nat Commun. 2022 Aug 20;13(1):4897. doi: 10.1038/s41467-022-32670-w. PMID 35986012
- [Background] Zhu Y, Mo M, Wei Y, Wu J, Pan J, Freedland SJ, Zheng Y, Ye D. Epidemiology and genomics of prostate cancer in Asian men. Nat Rev Urol. 2021 May;18(5):282-301. doi: 10.1038/s41585-021-00442-8. Epub 2021 Mar 10. PMID 33692499
- [Background] Wei Y, Wu J, Gu W, Qin X, Dai B, Lin G, Gan H, Freedland SJ, Zhu Y, Ye D. Germline DNA Repair Gene Mutation Landscape in Chinese Prostate Cancer Patients. Eur Urol. 2019 Sep;76(3):280-283. doi: 10.1016/j.eururo.2019.06.004. Epub 2019 Jun 24. PMID 31248605
- [Background] Gao D, Vela I, Sboner A, Iaquinta PJ, Karthaus WR, Gopalan A, Dowling C, Wanjala JN, Undvall EA, Arora VK, Wongvipat J, Kossai M, Ramazanoglu S, Barboza LP, Di W, Cao Z, Zhang QF, Sirota I, Ran L, MacDonald TY, Beltran H, Mosquera JM, Touijer KA, Scardino PT, Laudone VP, Curtis KR, Rathkopf DE, Morris MJ, Danila DC, Slovin SF, Solomon SB, Eastham JA, Chi P, Carver B, Rubin MA, Scher HI, Clevers H, Sawyers CL, Chen Y. Organoid cultures derived from patients with advanced prostate cancer. Cell. 2014 Sep 25;159(1):176-187. doi: 10.1016/j.cell.2014.08.016. Epub 2014 Sep 4. PMID 25201530
- [Background] Guo C, Figueiredo I, Gurel B, Neeb A, Seed G, Crespo M, Carreira S, Rekowski J, Buroni L, Welti J, Bogdan D, Gallagher L, Sharp A, Fenor de la Maza MD, Rescigno P, Westaby D, Chandran K, Riisnaes R, Ferreira A, Miranda S, Cali B, Alimonti A, Bressan S, Nguyen AHT, Shen MM, Hawley JE, Obradovic A, Drake CG, Bertan C, Baker C, Tunariu N, Yuan W, de Bono JS. B7-H3 as a Therapeutic Target in Advanced Prostate Cancer. Eur Urol. 2023 Mar;83(3):224-238. doi: 10.1016/j.eururo.2022.09.004. Epub 2022 Sep 13. PMID 36114082